CLINICAL TRIAL: NCT02378545
Title: (Feasibility) Open Label Randomised Controlled Trial of Hyperoxic O2 Therapy vs. Normoxic O2 Therapy in Sepsis
Brief Title: Trial of Hyperoxic O2 Therapy vs. Normoxic O2 Therapy in Sepsis
Acronym: HO2T or NO2T
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15/P/020; 2015-000629-35 (EudraCT Number)
Record Dates: First submitted 2015-02-12; First posted 2015-03-04 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2016-10

CONDITIONS: Sepsis
Keywords: Sepsis; Hyperoxia; Sepsis Six; Oxygen delivery
MeSH Terms: conditions — Sepsis; Hyperoxia | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyperoxia (Active Comparator): Oxygen will be administered using a non-re-breathe oxygen mask applied over the face and nose. The oxygen delivery device will be set to deliver oxygen at 15 litres per minute. The oxygen will be continuously delivered throughout the patients stay in the Emergency Department.
  Interventions: Drug: Oxygen
- normoxia (Active Comparator): Oxygen will not be administered if a patient's oxygen saturations (as measured using a pulse oximeter) are less than 94%. If a patient's oxygen saturations are less than 94%, oxygen will be 'titrated' using a 'venturi' type oxygen delivery device to achieve target saturations of 94%. Following initial dynamic titration (to identify correct oxygen delivery level) the oxygen delivery device will be re-evaluated hourly during the patient's stay in the emergency department.
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — On the Hyperoxia arm: Oxygen will be administered using a non-re-breathe oxygen mask applied over the face and nose.
  On the Normoxia arm: In many cases oxygen will not be administered. If required the minimum percentage required to reach the target saturations will be administered. In a majority of cases this will be via a venturi mask.
  Other Names: Medical Oxygen

SUMMARY:
The motivation for this study comes from a desire to improve the mortality of patients with sepsis. Oxygen is cheap, readily available and is included in current United Kingdom Emergency Department guidelines, but it may also be harmful to patients with sepsis - it is important to know if this is the case.

This study is a pilot study to also assess the feasibility of delivering a larger adequately powered study.

DETAILED DESCRIPTION:
Currently there is no consensus on the use of oxygen therapy in sepsis resuscitation. Uncertainty exists as to whether increasing oxygen above physiological levels (hyperoxia) or maintaining physiological oxygen concentration (normoxia) confers the most benefit to patients. By indicating whether hyperoxia is beneficial or not, the study hopes to further increase the effectiveness of sepsis resuscitation.

In patients with sepsis there are convincing, coherent pathophysiological and evidence-based justifications which support both normoxia and hyperoxia.

Why normoxia may benefit patients with sepsis: Enhanced oxidative and nitrosative stress resulting from increased formation of reactive oxygen species (ROS) and reactive nitrogen species (RNS) occurs during sepsis and is assumed to have major importance during the development of shock-related hypotension, impairment of microcirculatory perfusion, mitochondrial dysfunction, and tissue injury. It is well established that increasing the inhaled fraction of inspired oxygen (FiO2) leads to an increase in ROS production. The negative effects of hyperoxia in humans have been well demonstrated in a number of pathological conditions including stroke, myocardial infarction and some lung diseases. The pathological processes behind each of these conditions is very different from that of sepsis.

In a small observational study (88 patients) in patients with sepsis, of the hyperoxic patients, 8% died in hospital versus 6% with normoxia. Further prospective controlled trials are required. The deleterious effects of hyperoxia have also been demonstrated in a rat model.

Why hyperoxia may benefit patients with sepsis: Underlying cellular hypoxia, which may be difficult to detect, has been suggested as a major cause of morbidity and mortality in sepsis - this may be reversed or attenuated by high flow oxygen.

Hyperoxia may reverse arterial hypotension and exert anti-inflammatory and antiapoptotic properties. The beneficial effects of hyperoxia have been demonstrated in rat and pig models through increased survival and reduced inflammation.

One study in rats showed the most benefit on survival from oxygen administration when oxygen was administered in the first 4 hours of the trial, with no additional benefit beyond this time.

A further study (also in rats) demonstrated that 6 hours of oxygen per 24 hours for the first 48 hours following introduction of sepsis had the most beneficial anti-inflammatory effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or above.
* Diagnosed with presumed 'Sepsis'.
* Arrive at Derriford Emergency Department by ambulance.
* Provision of informed consent.
* Willing to allow their General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Female participants who are pregnant
* Existing diagnosis of chronic obstructive pulmonary disease (COPD)
* A primary diagnosis (or suspected diagnosis) of:

  * an acute cerebral vascular event
  * acute coronary syndrome
  * acute pulmonary oedema
  * status asthmatic
  * major cardiac arrhythmia (as part of primary diagnosis)
  * seizure
  * drug overdose
  * injury from burn or trauma
* Participants who require immediate intubation and ventilation on arrival in the Emergency Department
* Participants undergoing or have undergone cardiopulmonary resuscitation in the pre-hospital phase of their treatment.
* Current participation in another Clinical Trial of an Investigational Medicinal Product (CTIMP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-11-10 (Actual)

PRIMARY OUTCOMES:
Does delivery of high flow oxygen (hyperoxic oxygen therapy) compared to titrated oxygen therapy (normoxic oxygen therapy) reduce mortality at 90 days | 90 days
  Adult patients with sepsis presenting to the emergency department by ambulance.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Nutbeam, MBBS, Principal Investigator — University Hospital Plymouth NHS Trust
Locations (1):
- Plymouth Hospitals NHS Trust, Plymouth, Devon, United Kingdom